CLINICAL TRIAL: NCT05814224
Title: Monitoring luminAl Breast Cancer Through the Evaluation of Mutational and epiGeNEtic alteraTIons of Circulating ESR1 DNA
Acronym: MAGNETIC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2018.016
Record Dates: First submitted 2023-03-24; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Hormone Receptor Positive Breast Carcinoma; Breast Neoplasms; Neoplasms, Breast; Breast Diseases; Antineoplastic Agents; Aromatase Inhibitors; ESR1 Gene Mutation
Keywords: Epigenetics; Liquid biopsy; ctDNA; ESR1 Gene Mutation; Biomarker; HR-positive HER2-negative; Advanced breast cancer; CDK4/6; Antineoplastic Agents Hormonal
MeSH Terms: conditions — Breast Neoplasms; Breast Diseases | interventions — Liquid Biopsy; Tomography, X-Ray Computed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hormone-receptor positive MBC (Experimental): Women with hormone receptor-positive MBC, that will be eligible for endocrine therapy as first line treatment
  Interventions: Diagnostic Test: Liquid biopsy and CT scan

INTERVENTIONS:
Diagnostic Test: Liquid biopsy and CT scan — CT scan and liquid biopsy blood sample are performed at baseline, after 8 weeks from baseline and, then, every 12 weeks.
  Between two subsequent CT scan another liquid biopsy blood sample is performed.
  CEA and CA 15.3 will be performed at baseline and then concomitantly to the radiological evaluation

SUMMARY:
The purpose of the study is to determine the diagnostic role of ctDNA when used to monitor metastatic breast cancer (MBC) during first-line endocrine therapy.

DETAILED DESCRIPTION:
Patients with hormone receptor-positive MBC are eligible for endocrine therapy (ET) as first line treatment which is based on strategies aimed to either block signaling pathways depending on the estrogen receptor (ESR1) or using ESR1 antagonists. Only a few accepted predictive factors are associated with treatment benefit for MBC (i.e., hormone receptor status and HER2 status). Furthermore, a standardized assessment evaluation for MBC is still lacking. Because of these unmet needs, ET is continued until disease progression, or if toxicity requiring discontinuation occurs. Resistance is frequent in the treatment of early BC and unavoidable in MBC. Recently, mutations in ESR1 have been described in MBC that had been previously exposed to aromatase inhibitors (AIs) and are rarely detectable in primary BC. Besides that, resistance phenomena have been also linked to ESR1 cisregulatory elements (CRE, i.e. enhancers and promoters) hypermethylation, both related to ESR1 silencing.

According to the literature, the aim of the study is to detect tumor response with liquid biopsy technique compared to conventional clinical pratice algorithms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of adenocarcinoma of the breast with evidence of metastatic disease.
* ER positive tumor ≥ 1%
* HER2 negative breast cancer by FISH or IHC (IHC 0,1+, 2+ and/or FISH HER2: CEP17 ratio < 2.0)
* Females, 18 years of age or older
* Candidate to first-line endocrine therapy (LH-RH analogue for premenopausal women is allowed)
* Signed and dated informed consent document indicating that the subject (or legally acceptable representative) has been informed of all the pertinent aspects of the trial prior to enrollment.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Diagnosis of any secondary malignancy within the last 3 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix.
* Prior endocrine therapy for metastatic disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, 18 years of age or older
Enrollment: 164 (Estimated)
Dates: Start 2018-05-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Liquid-biopsy in monitoring treatment response in luminal breast cancer | 3 years
  The primary objective of this study is to evaluate whether liquid-biopsy technique is able to detect treatment response in luminal breast cancer through the quantification of ESR1 ctDNA mutations

SECONDARY OUTCOMES:
ctDNA/miRNA based follow-up | 3 years
  To characterize the clinical implications of deploying a ctDNA/miRNA based follow-up both in terms of outcome and health systems management.
Treatment resistance mechanisms | 3 years
  To investigate treatment resistance mechanisms and their detectability through ctDNA/miRNA analysis.
Specificity | From baseline until disease progression
  The proportion of patients correctly classified with a stable or response disease through the genetic and epigenetic analysis of ESR1 ctDNA among those without clinicoradiological relapse.
Positive predictive value | 3 years
  The proportion of patients correctly classified with a progressive disease through the genetic and epigenetic analysis of ESR1 ctDNA (i.e. those patients with molecular progression that is confirmed by clinic-radiological progression) among all patients with molecular progression (i.e. patients who show molecular progression irrespectively of clinic-radiological progression).
Negative predictive value | 3 years
  The proportion of patients correctly classified with a stable or response among those without clinico-radiological relapse.
Accuracy | 6 months
  Accuracy of the ESR1 ctDNA test in respect to correctly classify the patients with clinicoradiological relapse and without clinico-radiological relapse at 6 months.
Lead time (for PFS) | 3 years
  The time elapsed between the molecular detected progression and the imaging assessed one.
Number of futile diagnostic imaging | 3 years
  The number of imaging evaluations negative for progression and that could be avoided with the liquid biopsy technique.
Time to Progression (TTP) | 3 years
  The time from first biomarker assessment until objective tumor progression.
Progression Free Survival (PFS) | 3 years
  The time from first biomarker assessment until objective tumor progression or death for any cause, whichever comes first.
Overall Survival (OS) | 3 years
  The time from first biomarker assessment until death from any cause.
Overall Response Rate (ORR) | 3 years
  The sum of partial responses (PR) and complete responses (CR) evaluated from the time of first biomarker assessment to documented disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Puglisi, MD, Principal Investigator — Centro di Riferimento Oncologico - Aviano
Locations (7):
- Italy (7):
  - Asst Papa Giovanni Xxiii- Bergamo, Bergamo, Bergamo
  - Centro di Riferimento Oncologico - Aviano, Aviano, Pordenone
  - Asst Ospedali Civili Di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Policlinico G. Rodolico- San Marco-Catania, Catania
  - Universita' Degli Studi Di Napoli Federico Ii, Napoli
  - azienda sanitaria universitaria friuli centrale- Udine, Udine
  - Ospedale San Bortolo- Azienda Ulss8 Berica, Vicenza

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonotto M, Gerratana L, Di Maio M, De Angelis C, Cinausero M, Moroso S, Milano M, Stanzione B, Gargiulo P, Iacono D, Minisini AM, Mansutti M, Fasola G, De Placido S, Arpino G, Puglisi F. Chemotherapy versus endocrine therapy as first-line treatment in patients with luminal-like HER2-negative metastatic breast cancer: A propensity score analysis. Breast. 2017 Feb;31:114-120. doi: 10.1016/j.breast.2016.10.021. Epub 2016 Nov 9. PMID 27837704
- [Background] Toy W, Shen Y, Won H, Green B, Sakr RA, Will M, Li Z, Gala K, Fanning S, King TA, Hudis C, Chen D, Taran T, Hortobagyi G, Greene G, Berger M, Baselga J, Chandarlapaty S. ESR1 ligand-binding domain mutations in hormone-resistant breast cancer. Nat Genet. 2013 Dec;45(12):1439-45. doi: 10.1038/ng.2822. Epub 2013 Nov 3. PMID 24185512
- [Background] Jeselsohn R, Yelensky R, Buchwalter G, Frampton G, Meric-Bernstam F, Gonzalez-Angulo AM, Ferrer-Lozano J, Perez-Fidalgo JA, Cristofanilli M, Gomez H, Arteaga CL, Giltnane J, Balko JM, Cronin MT, Jarosz M, Sun J, Hawryluk M, Lipson D, Otto G, Ross JS, Dvir A, Soussan-Gutman L, Wolf I, Rubinek T, Gilmore L, Schnitt S, Come SE, Pusztai L, Stephens P, Brown M, Miller VA. Emergence of constitutively active estrogen receptor-alpha mutations in pretreated advanced estrogen receptor-positive breast cancer. Clin Cancer Res. 2014 Apr 1;20(7):1757-1767. doi: 10.1158/1078-0432.CCR-13-2332. Epub 2014 Jan 7. PMID 24398047
- [Background] Schiavon G, Hrebien S, Garcia-Murillas I, Cutts RJ, Pearson A, Tarazona N, Fenwick K, Kozarewa I, Lopez-Knowles E, Ribas R, Nerurkar A, Osin P, Chandarlapaty S, Martin LA, Dowsett M, Smith IE, Turner NC. Analysis of ESR1 mutation in circulating tumor DNA demonstrates evolution during therapy for metastatic breast cancer. Sci Transl Med. 2015 Nov 11;7(313):313ra182. doi: 10.1126/scitranslmed.aac7551. PMID 26560360
- [Background] Jansen MP, Martens JW, Helmijr JC, Beaufort CM, van Marion R, Krol NM, Monkhorst K, Trapman-Jansen AM, Meijer-van Gelder ME, Weerts MJ, Ramirez-Ardila DE, Dubbink HJ, Foekens JA, Sleijfer S, Berns EM. Cell-free DNA mutations as biomarkers in breast cancer patients receiving tamoxifen. Oncotarget. 2016 Jul 12;7(28):43412-43418. doi: 10.18632/oncotarget.9727. PMID 27270325
- [Background] Sasaki M, Tanaka Y, Perinchery G, Dharia A, Kotcherguina I, Fujimoto Si, Dahiya R. Methylation and inactivation of estrogen, progesterone, and androgen receptors in prostate cancer. J Natl Cancer Inst. 2002 Mar 6;94(5):384-90. doi: 10.1093/jnci/94.5.384. PMID 11880477
- [Background] Martinez-Galan J, Torres-Torres B, Nunez MI, Lopez-Penalver J, Del Moral R, Ruiz De Almodovar JM, Menjon S, Concha A, Chamorro C, Rios S, Delgado JR. ESR1 gene promoter region methylation in free circulating DNA and its correlation with estrogen receptor protein expression in tumor tissue in breast cancer patients. BMC Cancer. 2014 Feb 4;14:59. doi: 10.1186/1471-2407-14-59. PMID 24495356
- [Background] Stone A, Zotenko E, Locke WJ, Korbie D, Millar EK, Pidsley R, Stirzaker C, Graham P, Trau M, Musgrove EA, Nicholson RI, Gee JM, Clark SJ. DNA methylation of oestrogen-regulated enhancers defines endocrine sensitivity in breast cancer. Nat Commun. 2015 Jul 14;6:7758. doi: 10.1038/ncomms8758. PMID 26169690
- [Background] Panageas KS, Ben-Porat L, Dickler MN, Chapman PB, Schrag D. When you look matters: the effect of assessment schedule on progression-free survival. J Natl Cancer Inst. 2007 Mar 21;99(6):428-32. doi: 10.1093/jnci/djk091. PMID 17374832
- [Background] Bonotto M, Gerratana L, Poletto E, Driol P, Giangreco M, Russo S, Minisini AM, Andreetta C, Mansutti M, Pisa FE, Fasola G, Puglisi F. Measures of outcome in metastatic breast cancer: insights from a real-world scenario. Oncologist. 2014 Jun;19(6):608-15. doi: 10.1634/theoncologist.2014-0002. Epub 2014 May 2. PMID 24794159
- [Background] Bonotto M, Gerratana L, Iacono D, Minisini AM, Rihawi K, Fasola G, Puglisi F. Treatment of Metastatic Breast Cancer in a Real-World Scenario: Is Progression-Free Survival With First Line Predictive of Benefit From Second and Later Lines? Oncologist. 2015 Jul;20(7):719-24. doi: 10.1634/theoncologist.2015-0002. Epub 2015 May 27. PMID 26018662
- [Background] Fribbens C, O'Leary B, Kilburn L, Hrebien S, Garcia-Murillas I, Beaney M, Cristofanilli M, Andre F, Loi S, Loibl S, Jiang J, Bartlett CH, Koehler M, Dowsett M, Bliss JM, Johnston SR, Turner NC. Plasma ESR1 Mutations and the Treatment of Estrogen Receptor-Positive Advanced Breast Cancer. J Clin Oncol. 2016 Sep 1;34(25):2961-8. doi: 10.1200/JCO.2016.67.3061. Epub 2016 Jun 6. PMID 27269946
- [Background] Manavalan TT, Teng Y, Appana SN, Datta S, Kalbfleisch TS, Li Y, Klinge CM. Differential expression of microRNA expression in tamoxifen-sensitive MCF-7 versus tamoxifen-resistant LY2 human breast cancer cells. Cancer Lett. 2011 Dec 26;313(1):26-43. doi: 10.1016/j.canlet.2011.08.018. Epub 2011 Sep 10. PMID 21955614
- [Background] Miller TE, Ghoshal K, Ramaswamy B, Roy S, Datta J, Shapiro CL, Jacob S, Majumder S. MicroRNA-221/222 confers tamoxifen resistance in breast cancer by targeting p27Kip1. J Biol Chem. 2008 Oct 31;283(44):29897-903. doi: 10.1074/jbc.M804612200. Epub 2008 Aug 15. PMID 18708351